CLINICAL TRIAL: NCT03860571
Title: A Randomized, Placebo-Controlled, Sequential Single and Multiple Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral BT-11 in Healthy Adult Male and Female Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of Oral BT-11 in Healthy Adult Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-11-1a
Record Dates: First submitted 2019-02-03; First posted 2019-03-04 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Normal Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Simple randomisation using a randomisation table created by computer software (i.e. computerised sequence generation)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded:
  The people receiving the treatment/s The people administering the treatment/s The people assessing the outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BT-11 (Experimental)
  Interventions: Drug: BT-11

INTERVENTIONS:
Drug: Placebo — Oral tablet
  Arms: Placebo
Drug: BT-11 — Oral tablet
  Arms: BT-11

SUMMARY:
Study type: Interventional Description of intervention(s) / exposure

For single ascending dose, five dose target ranges of BT-11 (depending on body weight the doses in each cohort will be 5.9 - 7.7 mg/kg; 18.9 - 25.0 mg/kg; 44.3 - 50.0 mg/kg; 68.5 - 75 mg/kg and 94.2 - 100.0 mg/kg) will be evaluated, based on subject's weight on Day 1.

For multiple ascending dose (once daily for 7 days), three dose target ranges of BT-11 (depending on body weight the doses in each cohort will be 5.9 - 7.7 mg/kg; 44.3 - 50.0 mg/kg; and 94.2 - 100.0 mg/kg) will be evaluated, based on subject's weight on Day 1.

White tablets containing 500 mg BT-11 or matching placebo tablets will be dispensed.

Single ascending dose duration of administration will be once. For multiple ascending dose it will be up to 7 days.

The mode administration will be oral tablet. Compliance and adherence to the intervention will be performed based on the tablet return, tablet not consumed by the subject.

The safety monitoring committee will evaluate safety at conclusion of single ascending cohort 2 prior to the commencement of dosing for the multiple ascending dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male and female volunteers aged 18 to 65 years, inclusive.
2. Body weight 65 - 85 kg.
3. Volunteer has read, confirmed understanding of, and signed the written informed consent form after the nature of the study and all essential elements of the informed consent document have been fully explained and all of the Volunteer's questions have been answered to his or her satisfaction, prior to initiation of any study procedures.

Key Exclusion Criteria:

1. Any clinically significant abnormality identified in the screening history, physical examination (including Vital Signs), laboratory testing, or electrocardiographic testing. Repeat testing of vital signs to confirm the value is allowed. Up to two repeat tests are permitted to confirm eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 14 days

SECONDARY OUTCOMES:
PK | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Site, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No